CLINICAL TRIAL: NCT04724655
Title: Gastric Lavage With Paraffin Oil or Coconut Oil in Management of Acute Aluminum Phosphide Poisoning: A Randomized Controlled Clinical Trial.
Brief Title: Paraffin Oil or Coconut Oil in Acute Aluminum Phosphide Poisoning
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, samah maher, faculty of medicine,tanta university,Tanta Elgeesh street,qism 2,Egypt, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: oils and aluminum phosphide
Record Dates: First submitted 2021-01-19; First posted 2021-01-26 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Aluminum Phosphide Poisoning
MeSH Terms: interventions — Gastric Lavage; Mineral Oil; Bicarbonates; Coconut Oil; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- control group (Other): gastric lavage with saline and bicarbonate and standard treatment :inotropes as levophid, fluids and electrolytes , endotracheal intubation, mechanical ventilation and antiarrhythmic agents as Magnesium sulfate
  Interventions: Drug: standard treatment; Other: gastric lavage with saline and bicarbonate
- paraffin group (Active Comparator): gastric lavage with paraffin oil and bicarbonate and standard treatment :inotropes as levophid, fluids and electrolytes , endotracheal intubation, mechanical ventilation and antiarrhythmic agents as Magnesium sulfate
  Interventions: Other: gastric lavage with paraffin oil and bicarbonate; Drug: standard treatment
- coconut group (Active Comparator): gastric lavage with coconut oil and bicarbonate and standard treatment :inotropes as levophid, fluids and electrolytes , endotracheal intubation, mechanical ventilation and antiarrhythmic agents as Magnesium sulfate
  Interventions: Other: gastric lavage with coconut oil and bicarbonate; Drug: standard treatment

INTERVENTIONS:
Other: gastric lavage with paraffin oil and bicarbonate — Gastric lavage will be initiated with 50 mL of Paraffin oil and 50 mL of sodium bicarbonate solution 8.4%, then aspiration will be done after 3-5 min through nasogastric tube
  Arms: paraffin group
Other: gastric lavage with coconut oil and bicarbonate — Gastric lavage will be initiated with 50 ml coconut oil and 50 ml sodium bicarbonate 8.4 % then aspiration will be done after 3-5 min through nasogastric tube
  Arms: coconut group
Drug: standard treatment — inotropes as levophid, fluids and electrolytes , endotracheal intubation, mechanical ventilation and antiarrhythmic agents as Magnesium sulfate
Other: gastric lavage with saline and bicarbonate — Gastric lavage with saline and sodium bicarbonate 8.4% then aspiration will be done after 3-5 min through nasogastric tube
  Arms: control group

SUMMARY:
The aim of the present study is to evaluate safety and efficacy of gastric lavage with paraffin oil or gastric lavage with coconut oil in management of acute Aluminum phosphide poisoning.

DETAILED DESCRIPTION:
60 patients will be randomly assigned as control groups, paraffin group, and coconut group in a 1:1:1 ratio (30 patients in each group).

Inclusion criteria:

* Patients with symptomatic acute aluminum phosphide poisoning
* Age is more than 12 years of both gender
* Patients presenting within 6 hours post-ingestion of aluminum phosphide (Papade and Vanjari, 2019).

The diagnosis is made on the basis of:

1. The suggestive clinical manifestations due to and following shortly after a single exposure to aluminum phosphide.
2. Reliable identification of the compound based on the container brought by patient attendants.
3. Biochemical detection of phosphine gas in gastric aspirate (silver nitrate test).

   * Group (I): Gastric lavage with saline and sodium bicarbonate 8.4% then aspiration will be done after 3-5 min through nasogastric tube (Control group)
   * Group (II): Gastric lavage will be initiated with 50 mL of Paraffin oil and 50 mL of sodium bicarbonate solution 8.4%, then aspiration will be done after 3-5 min through nasogastric tube (Paraffin group).
   * Group (III): Gastric lavage will be initiated with 50 ml coconut oil and 50 ml sodium bicarbonate 8.4 % then aspiration will be done after 3-5 min through nasogastric tube (Coconut group).
   * All patients will continue to receive the standard supportive treatment according to Tanta University Poison Control Center protocol, which is determined by the attending physician who maintains clinical responsibility for all patients. Conventional standard treatment included using inotropes, fluids and electrolytes resuscitation, intubation, mechanical ventilation and antiarrhythmic agents if indicated.

ELIGIBILITY:
Inclusion Criteria:

* • Patients with symptomatic acute aluminum phosphide poisoning

  * Age is more than 12 years of both gender
  * Patients presenting within 6 hours post-ingestion of aluminum phosphide

Exclusion Criteria:

* • Patients less than 12 years of age

  * Pregnant and lactating women.
  * Patients with ingestion or exposure to other substances in addition to aluminum phosphide.
  * Patients with other major medical conditions (e.g. cardiovascular disease, diabetes mellitus, renal or hepatic failure).

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
death | 72 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Tantau, Tanta, Egypt